CLINICAL TRIAL: NCT05537467
Title: Effect of Music on Cardiopulmonary Exercise Capacity in Heart Failure Patients
Acronym: MUSIC-CPX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maya Ignaszewski (Other)
Responsible Party: Sponsor-Investigator, Maya Ignaszewski, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 76503
Record Dates: First submitted 2022-09-09; First posted 2022-09-13 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure
Keywords: Cardiopulmonary stress test; Exercise stress test; Cardiology; Exercise performance; Heart failure
MeSH Terms: conditions — Heart Failure | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music (Experimental): Music arm will listen to pre-selected music during their duration of the exercise testing via headphones that will be provided to the patients by the study personnel.
  Interventions: Other: Music
- Non-music (No Intervention): Non-music arm will not have pre-selected music playing during their duration of the exercise testing via the headphones provided to the patients by the study personnel.

INTERVENTIONS:
Other: Music — Patients randomized to the music group will listen to upbeat music using headphones.
  Arms: Music

SUMMARY:
The study aims to assess the effect of music on the heart resulting in a change in their exercise capacity among systolic heart failure patients undergoing Cardiopulmonary Exercise testing.

DETAILED DESCRIPTION:
Studies have previously shown the positive impact of music on the autonomic nervous system, neurohormonal and cardiovascular system. In addition, a previously published study found a positive impact of music resulting in an improvement of quality of life (QOL) in heart failure patients. Proposed mechanisms of benefit of music in heart failure include a reduction in sympathetic activity, and modulation of parasympathetic activity. Further, reduction in anxiety and arterial relaxation are thought to be beneficial effects of music. It is hypothesized that heart failure patients listening to music would have better exercise stress test performance and increased exercise time.

Adult patients with systolic heart failure scheduled to undergo Cardiopulmonary Exercise (CPX) testing at the Gill Heart and Vascular Institute will be recruited.

While the patients are undergoing Cardiopulmonary exercise testing, patients randomized to the 'music arm' will listen to pre-selected upbeat music during their duration of the exercise testing via headphones that will be provided to patients by the study personnel. The patients who are randomized to 'non-music arm' in which their headphones will not play music and the patients will perform the cardiopulmonary exercise testing as usual.

Standard clinical care is performing cardiopulmonary exercise testing without any music.

The investigators will then compare the results of CPX study of the two arms to assess the impact of music on exercise performance.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age >18 years)
* Able to consent
* English speaking

Exclusion Criteria:

* Severe hearing deficiency
* Unable to exercise.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-09-13 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Difference in O2 consumption (VO2) [L/min] | 15 minutes (at baseline 8 breaths, Anaerobic Threshold 8 breaths, Peak 8 Breaths)
  Assess above performance parameters in CPX and compare between Music and Non-Music arm.
Difference in CO2 production (VCO2) [L/min] | 15 minutes (at baseline 8 breaths, Anaerobic Threshold 8 breaths, Peak 8 Breaths)
  Assess above performance parameters in CPX and compare between Music and Non-Music arm.
Difference in respiratory exchange ratio (RER) | 15 minutes (at baseline 8 breaths, Anaerobic Threshold 8 breaths, Peak 8 Breaths)
  Assess above performance parameters in CPX and compare between Music and Non-Music arm.
Difference in Minute Ventilation (VE) [L/min] | 15 minutes (at baseline 8 breaths, Anaerobic Threshold 8 breaths, Peak 8 Breaths)
  Assess above performance parameters in CPX and compare between Music and Non-Music arm
Difference in Ventilatory Threshold (VT) [L] | 15 minutes (at baseline 8 breaths, Anaerobic Threshold 8 breaths, Peak 8 Breaths)
  Assess above performance parameters in CPX and compare between Music and Non-Music arm
Difference in respiratory rate (RR) [Breaths per minute] | 15 minutes (at baseline 8 breaths, Anaerobic Threshold 8 breaths, Peak 8 Breaths)
  Assess above performance parameters in CPX and compare between Music and Non-Music arm
Difference in Ventilatory Equivalent of CO2 (VE/VCO2) | 15 minutes (at baseline 8 breaths, Anaerobic Threshold 8 breaths, Peak 8 Breaths)
  Assess above performance parameters in CPX and compare between Music and Non-Music arm

SECONDARY OUTCOMES:
Difference in Heart Rate [Beats per minute] | 15 minutes (at baseline 8 breaths, Anaerobic Threshold 8 breaths, Peak 8 Breaths)
  Assess above performance parameters in CPX and compare between Music and Non-Music arm
Difference in O2 Pulse [ml] | 15 minutes (at baseline 8 breaths, Anaerobic Threshold 8 breaths, Peak 8 Breaths)
  Assess above performance parameters in CPX and compare between Music and Non-Music arm
Difference in Systolic and Diastolic Blood Pressure [mmHg] | 15 minutes (at baseline 8 breaths, Anaerobic Threshold 8 breaths, Peak 8 Breaths)
  Assess above performance parameters in CPX and compare between Music and Non-Music arm
Difference in Exercise time [mm:ss] | 15 minutes (Start to end of CPX study)
  Compare the CPX parameter between Music and Non-Music Arm
Difference in Work rate [watt] | 15 minutes (Start to end of each CPX study)
  Compare the CPX parameter between Music and Non-Music Arm

CONTACTS AND LOCATIONS:
Overall Officials: Maya T Ignaszewski, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No